CLINICAL TRIAL: NCT01836224
Title: A Prospective Open Label Randomized Non Inferiority Trial to Compare the Efficacy and Safety of Monotherapy With Noradrenaline and Terlipressin in Patients of Cirrhosis With Septic Shock Admitted to Intensive Care Unit.
Brief Title: Efficacy and Safety of Monotherapy With Noradrenaline and Terlipressin in Patients of Cirrhosis With Septic Shock Admitted to Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Sepsis-01
Record Dates: First submitted 2013-04-02; First posted 2013-04-19 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2013-12

CONDITIONS: Cirrhosis With Septic Shock
MeSH Terms: interventions — Terlipressin; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Noradrenaline (Active Comparator): Noradrenaline: Noradrenaline 2amp (4000mcg in 50ml) at 6ml/hr = 7.5mcg/min and dose maximum 60mcg/min 24ml/hr double strength. The dose to be increased every 15min from start dose by 1ml and to decrease by 0.5ml every 15min keeping MAP (Mean Arterial Pressure)>65.
  Interventions: Drug: Noradrenaline
- Terlipressin (Experimental): Terlipressin (1.3mcg/min i.e 2mg over 24 hr to max of terlipressin 5.2mcg/min i.e. up to 8mg over 24hr) .The dose to be increased every 15min from start dose by 1ml and to decrease by 0.5ml every 15min keeping MAP (Mean Arterial Pressure)>65 .Terlipressin 2mg in 48ml,1ml=42mcg=0.67mg/min, max dose 8mg/day- 8ml/hr of infusion.
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin — Terlipressin (1.3mcg/min i.e 2mg over 24 hr to max of terlipressin 5.2mcg/min i.e. up to 8mg over 24hr) .The dose to be increased every 15min from start dose by 1ml and to decrease by 0.5ml every 15min keeping MAP (Mean Arterial Pressure) >65 .Terlipressin 2mg in 48ml,1ml=42mcg=0.67mg/min, max dose 8mg/day- 8ml/hr of infusion.
  Arms: Terlipressin
Drug: Noradrenaline — Noradrenaline 2amp (4000mcg in 50ml) at 6ml/hr = 7.5mcg/min and dose maximum 60mcg/min 24ml/hr double strength. The dose to be increased every 15min from start dose by 1ml and to decrease by 0.5ml every 15min keeping MAP (Mean Arterial Pressure)>65
  Arms: Noradrenaline

SUMMARY:
The Patient evaluated in Emergency room since admission and detailed history and clinical examination done .The in hospital cases where sepsis is the culprit and shifted to Intensive Care Unit (ICU) in view of septic shock were included since onset of shock.

Initial fluid resuscitation done and if the patient were no fluid responsive they were randomized into arms noradrenaline or terlipressin and the dose escalated to achieve the primary objectives. At the same time the strict vitals monitoring and standard medical therapy for sepsis including antibiotics and other supportive therapy continued. The patients were followed up till discharge, death or up to 28days after enrollment into the protocol (whichever the longest). The detail methodology has been explained in column 14 later.

ELIGIBILITY:
Inclusion Criteria:

* Patient of cirrhosis or ACLF (Acute on Chronic Liver Failure) with septic shock (defined later).
* Age 18-70yrs
* An informed consent from the patient or relative

Exclusion Criteria:

* Pronounced cardiac dysfunction( valvular heart disease, coronary artery disease),
* Acute mesenteric ischemia (confirmed or suspected) or vasospastic diathesis (e.g. Reynaud's syndrome or related diseases).
* Pregnancy
* Previous history of transplantation on immunosuppressant.
* Acute gastrointestinal bleed.(defined later)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The Hemodynamic improvement as defined as mean arterial pressure > 65 mmHg. | 48 hrs

SECONDARY OUTCOMES:
Mortality | Day 3, Day 7 and Day 28
Number of organ system involved as defined by SOFA (Sequential Organ Failure Assessment) | Within 28 days
Days free of vasopressors | Within 28 days
Days free of ventilatory support | Within 28 days
Days free of steroid | Within 28 dyas
Length of stay | Within 28 days
Incidence of serious adverse events. | Within 28 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Choudhury A, Kedarisetty CK, Vashishtha C, Saini D, Kumar S, Maiwall R, Sharma MK, Bhadoria AS, Kumar G, Joshi YK, Sarin SK. A randomized trial comparing terlipressin and noradrenaline in patients with cirrhosis and septic shock. Liver Int. 2017 Apr;37(4):552-561. doi: 10.1111/liv.13252. Epub 2016 Oct 20. PMID 27633962